CLINICAL TRIAL: NCT03556683
Title: Phase I Assessment of Hypertonic Saline in Moderate to Severe Asthmatics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 17-3209; 17-0973 (Other: UNC RAMSES Number); 2P01HL108808-06 (NIH)
Record Dates: First submitted 2018-06-01; First posted 2018-06-14 (Actual); Results first posted 2025-05-04 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-05

CONDITIONS: Moderate to Severe Asthma
Keywords: asthma, hypertonic saline
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Intervention Model Description: To access the efficacy of inhalation of 3% and 7% hypertonic saline
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Early & Late-Phase Hypertonic Saline (HS) 7% (Cohort 1) (Experimental): Following screening, participants returned 1-6 weeks later and received albuterol alone followed by MCC. After another 1-6 weeks washout, participants then received late phase albuterol + 7% HS 4 hours post MCC. After another 1-6 weeks washout, participants then received albuterol + 7% HS followed by MCC. Five to ten days later participants returned for a discontinuation visit.
  Interventions: Device: 7% Hypertonic Saline; Drug: Salbutamol
- Hypertonic Saline (HS) 3% and 7% (Cohort 2) (Experimental): Following screening, participants returned 1-6 weeks later and received albuterol plus 3% HS followed by MCC. After another 1-6 weeks washout, participants then received albuterol + 7% HS followed by MCC. Five to ten days later participants returned for a discontinuation visit.
  Interventions: Device: 3% Hypertonic Saline; Device: 7% Hypertonic Saline; Drug: Salbutamol
- Acute Hypertonic Saline (HS) 7% (Cohort 3) (Experimental): Following screening, participants returned 1-6 weeks later and received albuterol alone followed by MCC. After another 1-6 weeks washout, participants then received albuterol + 7% HS followed by MCC. Five to ten days later participants returned for a discontinuation visit.
  Interventions: Device: 7% Hypertonic Saline; Drug: Salbutamol

INTERVENTIONS:
Device: 3% Hypertonic Saline — 4 mL of 3% hypertonic saline
  Arms: Hypertonic Saline (HS) 3% and 7% (Cohort 2)
Device: 7% Hypertonic Saline — 4 mL of 7% hypertonic saline
Drug: Salbutamol — 4 puffs (90 mcg/actuation)
  Other Names: Albuterol

SUMMARY:
Purpose: To determine if inhaled hypertonic saline (HS) accelerates airway mucociliary clearance (MCC) in well-controlled moderate to severe asthmatics.

DETAILED DESCRIPTION:
Participants: Non-smoking adults with well controlled moderate to severe asthma

Procedures (methods): After undergoing a general health screen, participants will undergo a lung transmission scan to create an image of the lungs. In subsequent visits, participants will inhale nebulized radiolabeled aerosol and sit in front of a gamma camera for 2 hours to measure clearance of radiolabeled particles from the lungs (procedure called gamma scintigraphy), which will be used to calculate baseline MCC. Spirometry will be performed before and at regular intervals after HS to assess for clinically significant reductions in lung function. Vital signs and symptom questionnaires will be administered as well. If participants are deemed tolerant to HS (i.e., no clinically significant deterioration in lung function, vital signs, or symptom questionnaire scores), participants will move forward with study visits.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 of both genders-
* Moderate to severe asthma at baseline (determined by Step 3 therapy or greater or by asthma impairment) and well-controlled asthma at the time of enrollment, as determined by NHLBI Expert Panel Report 3 guidelines for diagnosis and treatment of asthma.
* Negative pregnancy test for females who are not s/p hysterectomy with oophorectomy.
* Forced expiratory volume in 1 sec (FEV1) of at least 70% of predicted for age, sex, height, and race/ethnicity (without use of bronchodilating medications for 12 hours or long acting beta agonists for 24 hours).
* Documented COVID-19 vaccination

Exclusion Criteria:

Subjects who meet any of these criteria are not eligible for enrollment as study participants:

1. Clinical Contraindications:

   Any chronic medical condition considered by the PI as a contraindication to the study including significant cardiovascular disease, diabetes, chronic renal disease, chronic thyroid disease, history of chronic infections/immunodeficiency, or history of tuberculosis Any acute infection requiring antibiotics within 4 weeks of study. Mental illness or history of drug or alcohol abuse that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements.

   Medications which may impact the results of the study treatment, or may interfere with any other medications potentially used in the study (to include steroids, beta antagonists, non-steroidal anti-inflammatory agents) Active smoking to include e-cigarettes within 1 year of the study, or lifetime of > 10 pack-years of smoking Allergy/sensitivity to study drugs, or their formulations. History of intubation for asthma Unwillingness to use reliable contraception if sexually active (birth control pills/patch, condoms).

   Viral upper respiratory tract infection within 4 weeks of challenge. Radiation exposure history in the past year that would cause the participant to exceed Federal radiation safety guidelines.
2. Pregnant women and children (< 18 years as this is age of majority in NC) will also be excluded since the risks associated with hypertonic saline inhalation to the fetus or child and the risk of radiation are unknown and cannot be justified.
3. Use of the following medications:

   1. Systemic corticosteroids; subjects with systemic corticosteroid-dependent asthma will be excluded. All use of systemic steroids in the last year will be reviewed by a study physician.
   2. Use of daily theophylline within the past month
   3. Use of any immunosuppressant/immunomodulatory therapy within the preceding 12 months
   4. Use of beta blocking medications
   5. Receipt of Live Attenuated Influenza Vaccine (LAIV), also known as FluMist®, within the prior 30 days, or any vaccine within the prior 5 days
   6. Multivitamins, Vitamin C or E or herbal medications in the 4 days prior to the treatment visit
   7. Non-steroidal anti-inflammatory drugs in the 4 days prior to the treatment visit
   8. Subjects must be able to withhold morning doses of maintenance inhalers on the treatment days, including long acting bronchodilators and inhaled corticosteroids.
   9. Positive COVID-19 test in the prior 90 days.
4. Allergy/sensitivity to study drugs or their formulations: Known Immunoglobulin E (IgE) -mediated hypersensitivity to albuterol, diphenhydramine or corticosteroids.
5. Physical/laboratory indications:

   1. Abnormalities on lung auscultation
   2. Temperature > 37.8
   3. Systolic BP >150 mm Hg or < 90 mm Hg or diastolic BP> 90 mm Hg or < 50
   4. Oxygen saturation of < 93%
6. Inability or unwillingness of a participant to give written informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Peden, MD, MS, Principal Investigator — CEMALB
Locations (1):
- Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This exploratory study sought to determine the efficacy of 7% Hypertonic Saline (HS) for accelerating MCC acutely compared to baseline. Multiple cohorts evolved based on preliminary findings. Each cohort consisted of a Baseline MCC scan and albuterol+7% HS nebulization followed by MCC. In addition, differences in each cohort are as follows: cohort 1 late-phase 7% HS was assessed and in cohort 2, acute 3% HS was assessed and in cohort 3 acute albuterol alone was assessed.
Groups:
- Early & Late-Phase Hypertonic Saline (HS) 7% (Cohort 1): Following screening, participants returned 1-6 weeks later and received albuterol alone followed by MCC. After another 1-6 weeks washout, participants then received late phase albuterol + 7% HS 4 hours post MCC. After another 1-6 weeks washout, participants then received albuterol + 7% HS followed by MCC. Five to ten days later participants returned for a discontinuation visit.
  7% Hypertonic Saline: 4 mL of 7% hypertonic saline Salbutamol: 4 puffs (90 mcg/actuation), Albuterol
- Hypertonic Saline (HS) 3% and 7% (Cohort 2): Following screening, participants returned 1-6 weeks later and received albuterol plus 3% HS followed by MCC. After another 1-6 weeks washout, participants then received albuterol + 7% HS followed by MCC. Five to ten days later participants returned for a discontinuation visit.
  7% Hypertonic Saline: 4 mL of 7% hypertonic saline 3% Hypertonic Saline: 4 mL of 3% hypertonic saline Salbutamol: 4 puffs (90 mcg/actuation), Albuterol
- Acute Hypertonic Saline (HS) 7% (Cohort 3): Following screening, participants returned 1-6 weeks later and received albuterol alone followed by MCC. After another 1-6 weeks washout, participants then received albuterol + 7% HS followed by MCC. Five to ten days later participants returned for a discontinuation visit.
  7% Hypertonic Saline: 4 mL of 7% hypertonic saline Salbutamol: 4 puffs (90 mcg/actuation), Albuterol
Period: Overall Study
Arm/Group | Early & Late-Phase Hypertonic Saline (HS) 7% (Cohort 1) | Hypertonic Saline (HS) 3% and 7% (Cohort 2) | Acute Hypertonic Saline (HS) 7% (Cohort 3)
Started | 10 | 8 | 6
Completed | 9 | 7 | 6
Not Completed | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early & Late-Phase Hypertonic Saline (HS) 7% (Cohort 1) | Hypertonic Saline (HS) 3% and 7% (Cohort 2) | Acute Hypertonic Saline (HS) 7% (Cohort 3) | Total
Number analyzed (Participants) | 10 | 8 | 6 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 8 | 6 | 24
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 4 | 18
  Male | 1 | 3 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 9 | 8 | 6 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 3
  White | 8 | 7 | 4 | 19
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 8 | 6 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in MCC From Baseline to 7% Post Hypertonic Saline Inhalation
Description: This outcome was the primary outcome maintained across the entire study (all cohorts). Smaller cohorts also examined the effect of 7% HS on MCC 4 hours after inhalation (Cohort 1), the effect of 3% HS on MCC immediate inhalation (Cohort 2), and the effect of albuterol alone on MCC (Cohort 3).
Time Frame: Baseline MCC and at 2-12 weeks later MCC immediately after inhaled 7% HS, within approximately '15' minutes
Population: This outcome was the only outcome assessed across all cohorts of the study evaluating both the effect and tolerability of 7% HS immediately after inhalation. This is the most effective clinically relevant timepoint for effect and tolerability. For this endpoint, considering the entire sample size together was considered the most statistically sound way to report this outcome.
Measure: Mean (Standard Deviation); unit: percent clearance
Groups:
- Hypertonic Saline: Subjects will inhale hypertonic saline before having a Mucociliary Clearance (MCC) scan
  3% Hypertonic Saline: 4 mL of 3% hypertonic saline
  7% Hypertonic Saline: 4 mL of 7% hypertonic saline
Arm/Group | Hypertonic Saline
Number analyzed (Participants) | 22
percent clearance | 29.9 (7.9)
Statistical Analysis 1: Comparison: Hypertonic Saline; Effect immediately following hypertonic saline treatment; Test type: Superiority; p < 0.001, Mixed Models Analysis

2. Secondary Outcome: Effects of Hypertonic Saline on MCC by Testing
Description: The purpose of this outcome during Cohort 1 was to determine if there was a prolonged effect on MCC by 7% HS 4 hours post. Following interim analysis, it was decided that measurement at this timepoint would not be pursued and this outcome was deleted by a protocol amendment.
Time Frame: Baseline MCC, and 1-6 weeks later (MCC scan administered 4 hours after 7% HS inhalation)
Population: Only 9 participants underwent study for 4-hour effect of Hypertonic Saline which was only studied in Cohort 1.
Measure: Mean (Standard Deviation); unit: Percent clearance
Arm/Group | Early & Late-Phase Hypertonic Saline (HS) 7% (Cohort 1) | Hypertonic Saline (HS) 3% and 7% (Cohort 2) | Acute Hypertonic Saline (HS) 7% (Cohort 3)
Number analyzed (Participants) | 9 | 0 | 0
Percent clearance | 11.8 (8.3) |  |
Statistical Analysis 1: Comparison: Early & Late-Phase Hypertonic Saline (HS) 7% (Cohort 1); Effect of hypertonic saline 4 hours after treatment; Test type: Superiority; p = 0.99, Mixed Models Analysis

3. Secondary Outcome: The Proportion of Moderate to Severe Asthmatics Who Are Deemed 'Intolerant' to Hypertonic Saline
Description: A persistent reduction in the forced expiratory volume in one second (FEV1) of greater than or equal to 10% from that day's baseline
Time Frame: 30 minutes post-Hypertonic Saline
Population: This procedure was only done for Cohort 1. Data are reported for the 9 participants who completed the procedure.
Measure: Number; unit: proportion participants
Groups:
- Early & Late-Phase Hypertonic Saline (HS) 7% (Cohort 1): Following screening, participants returned 1-6 weeks later and received albuterol alone followed by MCC. After another 1-6 weeks washout, participants then received late phase albuterol + 7% HS 4 hours post MCC. After another 1-6 weeks washout, participants then received albuterol
- Hypertonic Saline (HS) 3% and 7% (Cohort 2): Following screening, participants returned 1-6 weeks later and received albuterol plus 3% HS followed by MCC. After another 1-6 weeks washout, participants then received albuterol + 7% HS followed by MCC. Five to ten days later participants returned for a discontinuation visit.
  7% Hypertonic Saline: 4 mL of 7% hypertonic saline 3% Hypertonic Saline: 4 mL of 3% hypertonic saline
Arm/Group | Early & Late-Phase Hypertonic Saline (HS) 7% (Cohort 1) | Hypertonic Saline (HS) 3% and 7% (Cohort 2) | Acute Hypertonic Saline (HS) 7% (Cohort 3)
Number analyzed (Participants) | 9 | 0 | 0
proportion participants | 0 |  |

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through study completion, up to approximately 3.5 months
Arm/Group | Early & Late-Phase Hypertonic Saline (HS) 7% (Cohort 1) | Hypertonic Saline (HS) 3% and 7% (Cohort 2) | Acute Hypertonic Saline (HS) 7% (Cohort 3)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 2/10 | 1/8 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early & Late-Phase Hypertonic Saline (HS) 7% (Cohort 1) (N=10) | Hypertonic Saline (HS) 3% and 7% (Cohort 2) (N=8) | Acute Hypertonic Saline (HS) 7% (Cohort 3) (N=6)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Mild Headache (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/83/NCT03556683/Prot_SAP_001.pdf
  • Informed Consent Form (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/83/NCT03556683/ICF_000.pdf